CLINICAL TRIAL: NCT07036653
Title: Bone Enhanced Ultrasound (BEUS) Data Library Development Project
Status: Not yet recruiting | Type: Observational
Sponsor: Queen's University (Other)
Responsible Party: Principal Investigator, Dr. Glenio Mizubuti (MD, PhD), Dr., Queen's University
Other Study IDs: 6043729
Record Dates: First submitted 2025-06-16; First posted 2025-06-25 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-06

CONDITIONS: Lower Back Pain; Facet Joint Pain; Low Back Pain; Osteoarthritis (OA)
Keywords: Facet joint injection; Spine ultrasound; 3D ultrasound; Low back pain
MeSH Terms: conditions — Low Back Pain; Osteoarthritis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: Individuals who have had a CT or MRI scans of their spine in the past 5 years
  Interventions: Diagnostic Test: spinal ultrasound

INTERVENTIONS:
Diagnostic Test: spinal ultrasound — Coronal, axial, sagittal scans of the spine using ultrasound

SUMMARY:
A common treatment for low back pain involves fluoroscopy-guided spinal facet joint injections and/or medial branch nerve blocks. Unfortunately, fluoroscopy requires expensive equipment and personnel and exposes patients and healthcare providers to ionizing radiation. Ultrasound offers a safer, lower-cost alternative, but the traditional 2-dimensional (2D) ultrasound systems are limited due to poor image quality, particularly in patients with higher body mass index (BMI).

As an alternative, a novel Bone Enhanced Ultrasound (BEUS) technology uses artificial intelligence (AI) to create real-time 3-dimensional (3D) images of the spine to guide needle placement for these injections. The AI software is trained by overlaying computed tomography (CT) and ultrasound images from a patient dataset to recognize anatomical landmarks. BEUS aims to ultimately replace fluoroscopy for spinal injections, reducing radiation exposure, lowering healthcare costs, and improving accessibility, especially in rural settings where CT and fluoroscopy are unavailable.

A key limitation, however, is that the current AI system is trained based primarily on patients (mostly pediatric) undergoing perioperative assessment of scoliosis. To address this, the current study aims to develop a new, more clinically relevant training AI dataset by collecting spinal ultrasounds from up to 100 adult participants (most/all of whom are followed at the local chronic pain clinic for low back pain) with existing spinal CT or magnetic resonance imaging (MRI) scans. This dataset will be used to retrain the current AI model to enhance the accuracy of 3D spinal reconstructions, thereby improving the clinical relevance of the BEUS system.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who have had previous CT or MRI scans of their spine in the past 5 years

Exclusion Criteria:

* < 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults who have had previous CT or MRI scans of their spine in the past 5 years
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Accuracy of 3D ultrasound spine reconstruction in adults with chronic low back pain | From enrollment to end of US scan (30 days)